CLINICAL TRIAL: NCT06331260
Title: Assessment of AFP and PIVKA-II as Prognostic Indicators in Liver Transplantation for Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Shulan (Hangzhou) Hospital (Other)
Responsible Party: Principal Investigator, Xiao Xu, Professor, Zhejiang University
Other Study IDs: CT2024-ZJU-OBS2
Record Dates: First submitted 2024-03-20; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Liver Transplantation; Hepatocellular Carcinoma; Alpha-Fetoprotein; Protein Induced by Vitamin K Absence or Antagonist-II
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preoperative AFP < 400 ng/mL or PIVKA-II < 200mAU/mL
- Preoperative AFP ≥ 400 ng/mL and PIVKA-II ≥ 200mAU/mL

SUMMARY:
As key biomarkers in HCC, AFP and PIVKA-II reflects biological features of tumor and has been widely applied for clinical diagnosis. Previous studies reported preoperative AFP and PIVKA-II are related to HCC recipient long-term survival after liver transplantation. However, there is no prospective study supporting these conclusions. This study aims to prospective collect liver transplantation cases from multiple transplant centers and further evaluate the prognostic role of preoperative AFP and PIVKA-II in liver transplantation for HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC based on CT or MRI imaging or needle biopsy confirming a histologic diagnosis of HCC.
2. Patients undergoing deceased donor liver transplantation for the first time.

Exclusion Criteria:

(1) patients who received split LT or simultaneous transplantation, (2) patients who received re-transplantation, (3) patients with macroscopic portal vein tumor thrombosis or other macrovascular invasion, (4) patients with incomplete follow-up, (5) taking warfarin at the time of LT biomarker measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients who undergoing deceased donor liver transplantation for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival rate | 2024.4.1-2028.4.1
Overall survival rate | 2024.4.1-2028.4.1
Tumor recurrence rate | 2024.4.1-2028.4.1